CLINICAL TRIAL: NCT02730676
Title: A Study to Assess Nicotine Pharmacokinetic Parameters of Digital Vapor Cigarettes in Adopters and Compare Them to Nicotine Pharmacokinetic Parameters of Cigarettes in Smokers
Brief Title: Comparison of Pharmacokinetic Parameters Between Adopters of Electronic Cigarettes and a Historical Sample of Combustible Cigarette Smokers
Status: Completed | Type: Observational
Sponsor: R.J. Reynolds Vapor Company (Industry)
Collaborators: Davita Clinical Research (Industry); RAI Services Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CSD1503
Record Dates: First submitted 2016-04-01; First posted 2016-04-06 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Smoking
Keywords: electronic cigarettes; e-cigarette; combustible cigarette; cigarette; menthol; cig-alike; subjective measures; pharmacokinetics; craving
MeSH Terms: conditions — Smoking; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, urine, buccal cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Electronic Cigarette #1: VUSE® Original Digital Vapor Cigarettes (29 mg nicotine)
  Interventions: Other: Electronic Cigarette #1
- Electronic Cigarette #2: VUSE® Menthol Digital Vapor Cigarettes (29 mg nicotine)
  Interventions: Other: Electronic Cigarette #2

INTERVENTIONS:
Other: Electronic Cigarette #1 — VUSE® Digital Vapor Cigarettes (original flavor, 29 mg nicotine)
  Other Names: VUSE® Original
  Groups: Electronic Cigarette #1
Other: Electronic Cigarette #2 — VUSE® Digital Vapor Cigarettes (menthol flavor, 29 mg nicotine)
  Other Names: VUSE® Menthol
  Groups: Electronic Cigarette #2

SUMMARY:
This study assesses the nicotine pharmacokinetic (PK) parameters in adopters of electronic cigarettes following a 12-hour tobacco and nicotine abstinence. The PK results of this study will be compared to historical data on smokers obtained in prior studies, as well as on naïve and short-term users of electronic cigarettes.

DETAILED DESCRIPTION:
This is an observational, open-label study to assess the nicotine pharmacokinetic (PK) parameters over a 6-hour period in adopters of electronic cigarettes with respect to an in-clinic 10-minute ad libitum period following a 12-hour tobacco and nicotine abstinence. In addition to PK parameters, subjective effects of urge for product will be assessed over a 6-hour period concurrently with the collection of the PK blood samples following a protocol defined schedule. The results of this study will be compared to historical PK and urge for product data obtained from smokers as well as naïve and short-term users of electronic cigarettes. In addition to the PK parameters and urge for product outcomes, plasma will be assessed for cotinine concentration prior to the 12-hour abstinence period.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English;
2. Generally healthy males and females, 21 to 60 years of age, inclusive, at Screening Visit;
3. Breath expired carbon monoxide (ECO) level is <10 parts per million (ppm) at the Screening Visit and Visit Day 1;
4. Positive urine cotinine test at the Screening Visit and Visit Day 1;
5. Electronic cigarettes are the only form of tobacco- or nicotine-containing product used within 30 days of Screening;
6. Willing to use VUSE digital vapor cigarettes during the study according to protocol;
7. Willing to be confined overnight and abstain from tobacco- and nicotine-containing product use for 12 hours prior to investigational product use through Study Discharge;
8. Females of childbearing age must be willing to use a form of contraception acceptable to the Investigator from the time of signing the ICF until Study Discharge, or be surgically sterile for at least 90 days prior to the Screening Visit;
9. Ability to safely perform study procedures, as determined by the Investigator;
10. Group 1-specific inclusion criteria includes the following:

    1. Currently uses VUSE Original digital vapor cigarettes;
    2. Self-reports using VUSE Original digital vapor cigarettes at least once daily, for at least one month prior to the Screening Visit.
11. Group 2-specific inclusion criteria includes the following:

    1. Currently uses VUSE Menthol digital vapor cigarettes;
    2. Self-reports using VUSE Menthol digital vapor cigarettes at least once daily, for at least one month prior to the Screening Visit.

Exclusion Criteria:

1. Presence of clinically significant or unstable/uncontrolled acute or chronic medical conditions at the Screening Visit, as determined by the Investigator, that would preclude a subject from participating safely in the study (e.g., uncontrolled hypertension, asthma or other lung disease, cardiac disease, neurological disease, or psychiatric disorders) based on safety assessments such as clinical laboratory tests, medical history, and physical/oral examinations;
2. Self-reports or safety labs indicate diabetes;
3. At risk for heart disease, as determined by the Investigator;
4. Use of medicine for treatment of depression or asthma;
5. Systolic blood pressure of ≥150 mmHg or a diastolic blood pressure of ≥95 mmHg, measured after being seated for 5 minutes;
6. Hemoglobin level <12 g/dL at the Screening Visit;
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus antibody (anti-HCV);
8. History or presence of hemophilia or other bleeding disorders;
9. History or presence of clotting disorders with concomitant use of anticoagulants;
10. Given a whole blood donation in the 8 weeks (≤56 days) prior to the Screening Visit;
11. Plasma donation within ≤7 days prior to the Screening Visit;
12. Body mass index <18.5 or >40.0 kg/m2 at the Screening Visit;
13. Weight of ≤110 pounds;
14. Poor peripheral venous access;
15. Postponing a decision to quit use of nicotine or tobacco products (defined as planning a quit attempt within 30 days of the Screening Visit) to participate in this study;
16. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within 30 days prior to the Screening Visit;
17. Females who test positive for pregnancy, are pregnant or breastfeeding, or plan to become pregnant during the course of the study;
18. A positive urine drug screen without disclosure of corresponding concomitant medication(s) at the Screening Visit or on Visit Day 1;
19. A positive alcohol breathalyzer result at Screening or on Visit Day 1;
20. Self-reports drinking more than 14 servings of alcoholic beverages per week (1 serving = 12 oz. of beer, 6 oz. of wine, or 1 oz. of liquor);
21. Participation in another clinical trial within 30 days prior to the Screening Visit, as determined from the last visit of the prior trial to the first Screening Visit in this study;
22. Employed by a tobacco or nicotine company, the study site, or handled tobacco or nicotine products as part of your job.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Generally healthy males and females 21 to 60 years of age who are exclusive users of electronic cigarettes.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine area under the plasma nicotine concentration versus time curve (AUC)
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine maximum plasma concentration (Cmax), baseline adjusted

OTHER OUTCOMES:
Nicotine pharmacokinetics with respect to initiation of in-clinic investigational product use following a 12-hour tobacco and nicotine abstinence | -5, -0.5, 5, 7.5, 10, 15, 20, 30, 45, 60, 75, 90, 120, 150, 180, 240, 300, 360 minutes
  Determine time to maximum plasma nicotine concentration (Tmax), baseline adjusted
Subjective effects scores for Urge for Product (UFP) with respect to initiation of in-clinic investigational product use following a 12-hour tobacco and nicotine abstinence | -30, 5, 15, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360 minutes
  Score subjective effects using a numeric rating scale to determine area under the UFP score-versus-time curve (AUEC)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Williams, MD, Principal Investigator — Davita Clinical Research
Locations (1):
- Davita Clinical Reserch, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No